CLINICAL TRIAL: NCT02618343
Title: A Randomized Control Equivalence Study of Emergency Medical Services Use of Isopropyl Alcohol Aromatherapy Versus Ondansetron for Treatment of Pre-hospital Nausea
Brief Title: EMS Use of Isopropyl Alcohol Aromatherapy Versus Ondansetron
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-859H
Record Dates: First submitted 2015-11-22; First posted 2015-12-01 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Nausea
MeSH Terms: conditions — Nausea | interventions — 2-Propanol; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- ISOPROPYL ALCOHOL AROMATHERAPY (Experimental): Prehospital patients complaining of nausea randomized into the IPA Arm.
  Interventions: Drug: IPA
- Ondansetron (Active Comparator): Prehospital patients complaining of nausea randomized into the ondansetron arm.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: IPA — IPA Aromatherapy for the experimental arm
  Other Names: rubbing alcohol
  Arms: ISOPROPYL ALCOHOL AROMATHERAPY
Drug: Ondansetron — Zofran will be administered to the Control arm. This is the drug historically administered by prehospital personnel.
  Other Names: Zofran
  Arms: Ondansetron

SUMMARY:
Nausea is a common symptom encountered in the Emergency Medical Services (EMS) environment that is often treated with oral or intravenous anti-emetic medications. Research Design/Plan: This will be a randomized equivalence study comparing the reduction in a patient's reported level of nausea after treatment with either Ondansetron or IPA Methods: Patients who report nausea and/or vomiting in the normal evaluation and care of after calling 911 for Emergency Medical Care will be offered enrollment in the study. A short script will be attached to the outside of each study packet providing information about the study and its risks and benefits. Verbal or written (waiver of informed consent will be requested) permission will be obtained to start randomization. If the patient agrees to enroll then the study packet will be opened and utilized. All Advanced Life Support Ambulances in the San Antonio Fire Department will have sealed numbered opaque boxes or envelopes with either: 70% Isopropyl Alcohol swabs or ondansetron. Six Visual Nausea Severity Scoring cards will be provided with a marking pen to record timed nausea levels before and upon arrival to the Emergency Department and 15 minutes after treatment whichever comes first.

Clinical Relevance: This treatment has not been studied in the unique environment encountered by Paramedics in the Pre-Hospital setting. If this treatment is found to be effective, it many offer a very simple, extremely inexpensive and non-invasive (basic life support) approach for the treatment of nausea.

DETAILED DESCRIPTION:
Nausea is a common symptom encountered in the Emergency Medical Services (EMS) environment that is often treated with oral or intravenous anti-emetic medications. Post operative patients with modern anesthesia techniques and processes still have a 20-30% incidence of Nausea and/or vomiting. Nausea is a complicated symptom that is though to arise from the vomiting center in the lateral reticular formation in the brainstem. Afferent inputs form the cerebellum, higher cortical centers, the vestibular apparatus, the glossopharyngeal nerve and the vagal nerve inputs contribute to the process of the perception of nausea. Chemoreceptors in the Chemoreceptor Trigger Zone (CTZ) are located on the brain surface and are highly vascularized leading to increased exposure to neurotransmitters such as Serotonin (5-HT-3), histamine (H1) acetylcholine and dopamine. Blocking such neurotransmitter stimulation with targeted medications such as antihistamines or 5-HT-3 antagonists such as Ondansetron.

Nausea is a common symptom encountered in the Emergency Medical Services (EMS) environment that is often treated with oral or intravenous anti-emetic medications. Many patients do not respond well to this therapy, and EMS services that have only basic life support (BLS) capabilities may not have any good treatment currently. Additionally, because of the configuration of modern day ambulances, the patient is transport in a rear facing position in the patient compartment with very limited view of the environment. This method of transport frequently causes motion sickness.

Motion sickness is thought to be caused by inadequate adaption of the body to conflicts between vestibular, visual, other proprioceptive inputs and inhibition of the vestibular cerebellum. Common therapies may include antihistamines, benzodiazepines, tricyclic antidepressants and or scopolamine. Behavioral strategies such a watching the true horizon, steering the vehicle, tilting head into turns and laying down with eyes closed have been shown to alleviate some symptoms of motion sickness. But these strategies are not available in the EMS environment. Scopolamine administered well before motion stimulus has been shown to prevent motion sickness and acute treatment is best when using sedating antihistamines. Non-sedating antihistamines, Ondansetron and ginger root have not been found to effectively prevent nor treat motion sickness.

Multiple agents have been studied for the treatment of nausea in the emergency department with equivalency of effect and time on onset. Common agents include ondansetron, metoclopramide, promethazine and prochlorperazine. Such agents have also been used in the EMS environment to some degree, but require parenteral administration with exposure to the risks for side effects or sedation. There are also not options at the BLS level. Post-operative oxygen therapy has not been shown to decrease post nausea after c-section delivery which is disappointing as this is a ubiquitous therapy in the EMS environment of care, is inexpensive and easy to administer. Ondansetron has been shown to be safe and effective in the prehospital environment with a low incidence of side effects but cost and need for parenteral administration is often a barrier to care.

Multiple studies have shown Isopropyl Alcohol (IPA) 70% aromatherapy to be as effective as Ondansetron with a more rapid onset of nausea relief. This therapy was performed by holding a folded saturated 70% IPA pad under the nares with the patient inhaling the vapors. The patient is simply instructed to take three deep breaths through their nose. In animal experiments, toxicity from inhalation of IPA is very low at doses allowable by inhalation as compared with dermal or oral ingestion. Dermal application of IPA is routinely used by EMS personnel to cleanse the area of skin immediately surrounding the insertion point of an intravascular catheter for medication administration, or blood draw.

PURPOSE:

IPA Therapy may offer a very inexpensive, easy to administer, and effective alternative to medication therapy for nausea and vomiting in the prehospital.

RECRUITMENT AND RANDOMIZATION PROCESS Patients who report nausea and/or vomiting in the normal evaluation and care of after calling 911 for Emergency Medical Care will be offered enrollment in the study.

A short script will be attached to the outside of each study packet providing information about the study and its risks and benefits. Verbal or written (waiver of informed consent will be requested) permission will be obtained to start randomization. If the patient agrees to enroll then the study packet will be opened and utilized.

PROCEDURES AND LOGISTICS

All Advanced Life Support Ambulances in the San Antonio Fire Department will have sealed numbered opaque boxes or envelopes with either:

* Three large 2 ply 70% Isopropyl Alcohol swabs OR
* Ondansetron (Zofran) 4mg for IV/IM use

These study packets will have similar weight, shape and contour despite the contents. If needed, props may be includes to make packages similar in weight, contour or sound when shaken so as to not reveal its true contents. The goal is to enroll at least 400 patients over a 1 year period.

For each arm, the package will contain a step by step instruction checklist. Six Visual Nausea Severity Scoring cards will be provided with a marking pen to record timed nausea levels before and upon arrival to the Emergency Department and 15 minutes after treatment whichever comes first. The treatment protocol for each arm will be:

70% Isopropyl Alcohol

1. Mark Time and Visual Nausea Severity Score 0-10
2. Remove alcohol prep with gloved hand
3. Place under nares of the patient
4. Instruct the patient to take three separate deep inhalations of the Isopropyl vapors through their nose
5. Record time of treatment on back of first Visual Nausea Severity Score card.
6. Mark time and Subsequent Visual Nausea Severity Scores upon arrival to the Emergency Department at indicated time intervals.
7. If patient still has significant nausea and or vomiting after ten minutes provide rescue Ondansetron therapy with 4mg of Ondansetron slow IV push or IM
8. Mark time and Visual Nausea Severity Score upon arrival to the Emergency Department on third card.
9. Document all interventions on electronic Patient Care record as per usual procedures.
10. Complete Paramedic evaluation tool.
11. Envelope or box, with Consent, score cards and Paramedic evaluation tool will be returned to Medic Officer on duty and a new study packet will be replaced.
12. Used Study Packets will be collected by the Investigators

Ondansetron 4mg IV/IM (standard of care)

1. Mark Time and Visual Nausea Severity Score 0-10 on first enclosed card.
2. Start IV if not already done so.
3. If unable to obtain IV access in two attempts use intramuscular route.
4. Inject 4mg of Ondansetron slow IV push or IM.
5. Record time of treatment on back of first Visual Nausea Severity Score card.
6. Mark time and Second Visual Nausea Severity Score upon arrival to the Emergency Department or 10 minutes after treatment whichever comes first.
7. If patient still has significant nausea and or vomiting after ten minutes provide rescue an additional dose of Ondansetron therapy with 4mg of Ondansetron slow IV push or IM
8. Mark time and Visual Nausea Severity Score upon arrival to the Emergency Department on third card.
9. Document all interventions on electronic Patient Care record as per usual procedures.
10. Complete Paramedic evaluation tool.
11. Envelope or box, with Consent, score cards and Paramedic evaluation tool will be returned to Medic Officer on duty and a new study packet will be replaced.
12. Used Study Packets will be collected by the Investigators.

Data Analysis Plan:

A secure excel spreadsheet tool will be used to abstract data from the research data collection documents and the EMS electronic patient care record. The patient will only be identified by the randomization number, incident number, age (if greater than 89 age will be indicated by <89 years), sex and date of service in the database and on all study packet materials. All relevant time intervals and Visual Nausea Severity Scores will be recorded for enrolled patients. Time to treatment will be compared between the two arms of the study as well as changes in Visual Nausea Severity Scores. Treatment failures requiring additional Ondansetron will be characterized. Paramedic will be asked to evaluate the treatment provided for ease of use, time needed to complete the treatment and their impression of effectiveness of the assigned treatment. T-test and confidence intervals will be utilized to determine statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Adults (non-pregnant) age 18 years or older with a symptom of nausea and/or vomiting requiring treatment by EMS

Exclusion Criteria:

* Children not yet 18 years of Age
* Prisoners or those under arrest
* Patients known or suspected to be Pregnant
* Clinical Intoxication
* Patients unable to provide informed consent
* Recent Upper respiratory Tract infection
* Inability to follow instructions
* Inability to inhale through Nares

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- San Antonio Fire Department EMS Division, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients being transported to the hospital by EMS will be recruited
Groups:
- Isopropyl Alcohol: Prehospital nausea patient randomized into the IPA group
- Ondansetron Group: Prehospital nausea patient randomized to the Ondansetron group
Period: Overall Study
Arm/Group | Isopropyl Alcohol | Ondansetron Group
Started | 28 | 23
Completed | 28 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ISOPROPYL ALCOHOL AROMATHERAPY | Ondansetron | Total
Number analyzed (Participants) | 28 | 23 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Age Data not collected | NA (NA) — Age Data not collected | NA (NA) — Age Data not collected
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — These data were not collected | NA — These data were not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — These data were not collected | NA — These data were not collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | NA — Race and Ethnicity Not Collected | NA — Race and Ethnicity Not Collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian | NA — Race and Ethnicity Not Collected | NA — Race and Ethnicity Not Collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | NA — Race and Ethnicity Not Collected | NA — Race and Ethnicity Not Collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | NA — Race and Ethnicity Not Collected | NA — Race and Ethnicity Not Collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | NA — Race and Ethnicity Not Collected | NA — Race and Ethnicity Not Collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race | NA — Race and Ethnicity Not Collected | NA — Race and Ethnicity Not Collected | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | NA — Race and Ethnicity Not Collected | NA — Race and Ethnicity Not Collected | NA — Total not calculated because data are not available (NA) in one or more arms.
Nausea level [Mean (Standard Deviation); unit: units on a scale] — The scale used was a 10 cm visual analog scale with 10 being severe nausea, and 0 being nausea free
  units on a scale | 4.3 (3.1) | 3.6 (2.9) | 4.0 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Time to Nausea Reduction by 50% by Visual Analog Scale.
Description: A visual analog scale (VAS) will be utilized to determine level of nausea. The VAS scale will be utilized before enrollment, at the time of medication administration, then every 2 minutes after administration for 10 minutes. The scale is a numbered linear scale from 0-10, with 0 = no nausea and 10 = worst nausea possible
Time Frame: Baseline and up to 10 minutes
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Isopropyl Alcohol | Ondansetron Group
Number analyzed (Participants) | 28 | 23
Minutes | 4.3 (3.1) | 3.5 (2.9)

2. Secondary Outcome: Number of Subjects That Required Rescue Ondansetron
Description: We will compare the number of times that a subject required ondansetron administration after IPA administration, and the number of times ondansetron repeat dose is required in the control group.
Time Frame: 15 minutes
Population: EMS Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Isopropyl Alcohol | Ondansetron Group
Number analyzed (Participants) | 23 | 28
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events are recorded from time of initial administration to 15 minutes after arrival at the emergency room. Duration varies according to length of time that it takes to transport the participant from pick up location to the emergency room.
Arm/Group | Isopropyl Alcohol | Ondansetron Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/23
Other Adverse Events (participants affected / at risk) | 0/28 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT02618343/Prot_SAP_000.pdf